CLINICAL TRIAL: NCT07197307
Title: Combining Loncastuximab Tesirine and Epcoritamab in Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: CLEAR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: AbbVie (Industry); Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WWU23_0006; 2023-509861-19-01 (EU CTIS Number)
Record Dates: First submitted 2025-09-03; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Aggressive Diffuse Large B-cell Lymphoma; High-grade B-cell Lymphoma (HGBL); Follicular Lymphoma (FL) Grade 3B
Keywords: Loncastuximab Tesirine; Epcoritamab; Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Loncastuximab Tesirine and Epcoritamab (Experimental): Combination of loncastuximab tesirine and epcoritamab in patients with relapsed/refractory aggressive B-cell lymphoma (DLBCL, HGBL or FL grade 3B)
  Interventions: Drug: Loncastuximab Tesirine and Epcoritamab

INTERVENTIONS:
Drug: Loncastuximab Tesirine and Epcoritamab — Combination therapy of loncastuximab tesirine and epcoritamab

SUMMARY:
This is a phase II study designed to evaluate the toxicity and efficacy of the combination of loncastuximab tesirine and epcoritamab in patients with relapsed/refractory aggressive B-cell lymphoma. Chimeric antigen receptor (CAR)-T cell naive patients who have failed first-line therapy and patients who have received CAR-T cells as second-line therapy and experienced CAR-T failure will be eligible for inclusion.

DETAILED DESCRIPTION:
A total of 120 patients will be included. 60 days after 20 patients have started the therapy, a safety analysis will be performed to identify early and unexpected side effects of the combination therapy. An interim analysis will be conducted 6 months after recruitment of the 50th patient to check the effectiveness of the therapy.

ELIGIBILITY:
Inclusion Criteria:

Disease:

1. Subjects with histologically confirmed relapsed/refractory DLBCL based on pathology report (WHO 2022 criteria)

   1. DLBCL (de novo or transformed)
   2. High-grade B-cell lymphoma with MYC and BCL2 rearrangements
   3. High-grade B-cell lymphoma, not otherwise specified (NOS)
   4. Follicular lymphoma grade 3B

   Diagnostic biopsy performed at the time of relapse/progressive disease no longer than 3 months before study entry must be available, with sufficient material for central review and complimentary scientific analyses. CD20 expression (or a high likelihood of CD20 expression) based on immunohistochemistry should be documented prior enrollment into the study.

   Refractory disease is defined as no remission to the last therapy. Subjects intolerant to previous therapy are excluded. Two groups of patients are eligible:
   * Progressive disease (PD) or stable disease (SD) as best response to previous therapy.
   * Complete (CR) or partial response (PR) as the best response after previous therapy, with biopsy-proven relapse occurring < 6 months after end of treatment.

   Relapsed disease is defined as subjects achieving complete or partial remission to previous therapy, followed by biopsy-proven relapse ≥6 months after treatment completion. Subjects with refractory and early relapsed (≤12 months) disease after first line anti-CD20-/anthracycline-containing therapy are eligible. Subjects with late relapsed (>12 months) disease after first line anti-CD20-/anthracycline-containing therapy can be enrolled in the study only if deemed ineligible to high dose chemotherapy (HDCT) followed by autologous stem cell transplantation (ASCT). Subjects relapsed/refractory to second line CAR-T cell therapy are eligible.
2. Subject must be 18 years or older.
3. Subject must be eligible to receive and in need of treatment initiation based on symptoms and/or disease burden, as assessed by the investigator.
4. Eastern Cooperative Oncology Group Performance (ECOG) status 0-2.
5. Subject must have one or more measurable disease sites defined as follows:

   1. A positron emission tomography/computed tomography (PET/CT) scan demonstrating PET- positive lesion(s) AND
   2. At least one measurable nodal lesion (long axis > 1.5 cm and short axis > 1.0 cm) or ≥ one measurable extra-nodal lesion (long axis > 1.0 cm) on CT scan or MRI.
6. Ability to understand and willingness to sign written informed consent. Signed informed consent must be obtained before any study specific procedure.

   Contraception:
7. Women of childbearing potential and sexually active men must practice a highly effective method of birth control during and after the study, consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men with female partners who are of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of giving informed consent until at least 7 months after the patient receives his last dose of study treatment. Men must agree not to donate sperm from the time of giving informed consent until at least 7 months after the patient receives his last dose of study treatment. For female subjects, they apply for 12 months after the last dose of the study drug. A woman is considered to be of childbearing potential until becoming post-menopausal or permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. Post-menopausal status is defined as no menstrual periods for a continuous 12-month period without an alternative medical cause. A post-menopausal state can be confirmed by a high follicle-stimulating hormone (FSH) level within the postmenopausal range, especially in women not using hormonal contraception or replacement therapy. The investigator or a designated associate will provide guidance to patients on achieving highly effective contraception (with a failure rate of less than 1%), such as intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, having a vasectomized partner, or sexual abstinence. Male patients are required to use condoms unless their female partner is permanently sterile.
8. Women of childbearing potential participating in the study will be required to undergo a pregnancy test using either urine or serum beta-human chorionic gonadotropin (beta-hCG) at the screening visit. A negative result is necessary for inclusion in the study.

   Adequate baseline organ function tests collected no more than 7 days before starting study treatment:
9. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), except for patients with Gilbert syndrome, cholestasis due to hepatic hilum adenopathies or liver involvement, or biliary obstruction due to lymphoma, who may have a total bilirubin ≤ 3 times the ULN.
10. Alanine transaminase (ALT) and aspartate aminotransferase (AST) and gamma-glutamyl transferase (GGT) ≤ 2.5 times the ULN, or ≤ 5 times the ULN for patients with liver involvement by lymphoma.
11. Glomerular filtration rate (GFR) ≥ 45 mL/min/1.73 m² according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. If not initially within target range, this evaluation may be repeated after at least 24 hours, either using the CKD-EPI formula or by 24-hour sampling. If the subsequent result is within the acceptable range, it may be used to fulfill the inclusion criteria.
12. Prothrombin time/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 times the ULN, unless the patient is receiving anticoagulation (although the INR should not exceed 4.0).
13. Platelet count ≥ 75,000/mm³ without transfusion in the prior 7 days.
14. Hemoglobin ≥ 8 g/dL.
15. Absolute neutrophil count ≥ 1,000/mm3 (off growth factors at least 72 hours).
16. Left ventricular ejection fraction > 45%.

    Concomitant Medications:
17. Subjects should not be taking any active medication known to decrease T-cell numbers or activity, or any other concurrent immunosuppressive medication, except for up to 10 mg of prednisone daily or an equivalent dose, unless it is necessary for disease control during the screening period, premedication and/or cytokine release syndrome (CRS)/ immune effector cell-associated neurotoxicity syndrome (ICANS) management within the study.
18. Subjects must not have been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of the study drug. They should not be currently enrolled in another interventional clinical study or have been previously enrolled in this study, unless the agent being used has been approved under emergency authorization (e.g., anti-severe acute respiratory syndrome coronavirus (SARS-CoV-2) monoclonal antibodies).
19. Acute toxicity (except alopecia, fatigue) of any prior lymphoma therapy should be resolved to Grade ≤ 1 (with the exception of prior CRS or ICANS that should be fully resolved) at study screening.
20. The subject should not have received vaccination with live-attenuated vaccines within 28 days prior to screening, and they should not be expected to require any live-attenuated vaccination during their participation in the study, including at least 3 months following the last dose of study treatment. However, vaccination with coronavirus messenger ribonucleic acid (mRNA) and adenovirus-based vaccines, which are not live-attenuated vaccines, is permitted.

Exclusion Criteria:

Patients who meet any of the following criteria at the time of screening will be excluded:

1. Any prior lymphoma-directed treatment, except for first-line anti-CD20-/anthracycline-containing chemoimmunotherapy or second line CAR-T cell therapy. Particularly, patients previously treated with loncastuximab tesirine and any CD3xCD20 bispecific antibody therapy are not eligible.
2. Patients with late relapse (>12 months) after first-line immunochemotherapy considered HDCT/ASCT eligible as assessed by the local investigator.
3. Known central nervous system (CNS) involvement.
4. Diagnosed or treated for any malignancy other than r/r DLBCL, HGBL or FL grade 3B within the last 3 years, except for adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, non-invasive basal cell or squamous cell skin carcinoma, adequately treated carcinoma in situ without evidence of disease, localized prostate cancer, post-radical prostatectomy with non-rising prostate-specific antigen levels < 0.1 ng/mL, cervical carcinoma of stage 1B or less, non-invasive, superficial bladder cancer or any curable cancer with a CR of > 2 years duration.
5. Known history of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or active hepatitis B virus (HBV) infection or any known active systemic bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds). Patients with serologic markers of HBV immunization due to vaccination (HBsAg negative, Anti-HBc negative, and Anti-HBs positive) will be eligible. Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
6. Cytomegalovirus (CMV)-PCR positive at baseline.
7. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or interfere with the feasibility to administer study drugs including active hemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS), history of cutaneous collagenous vasculopathy and capillary leak syndrome.
8. Concurrent treatment with another investigational agent or radiation therapy.
9. Any psychological, cognitive, familial, or social condition that, in the investigator's opinion, compromises the patient's ability to understand the patient information, give informed consent, or comply with the study protocol.
10. Participation in another clinical trial.
11. Known history of hypersensitivity and/or positive serum human anti-drug antibody (ADA) against any component of the study products or of the concomintant medication or an anti-CD19 antibody.
12. History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
13. Clinically significant third space fluid accumulation, such as ascites requiring drainage or pleural effusion that either requires drainage or is associated with shortness of breath.
14. Pregnancy or breastfeeding.
15. Use of any other experimental medication within 30 days or 5 half-lives prior to the start of the study drug (Cycle 1 Day 1).
16. Close affiliation with the investigational site, such as being a close relative of the investigator or dependent person (e.g., employee or student of the investigational site).

    Excluded medical conditions:
17. Congestive heart failure > New York Heart Association (NYHA) class 2.
18. Unstable angina (angina symptoms at rest) or new-onset angina (begun within the last 3 months).
19. Uncontrolled atrial or ventricular cardiac arrhythmia.
20. Left ventricular ejection fraction ≤ 45%.
21. Electrocardiographic evidence of acute ischemia, coronary angioplasty, or myocardial infarction within 6 months prior to screening.
22. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 3 months before the start of study medication.
23. Congenital long QT syndrome or a QT corrected by Fridericia's formula (QTcF) interval of > 480 ms at screening (unless secondary to pacemaker or bundle branch block).
24. Severe chronic pulmonary disease.
25. Known clinically significant liver disease, including hepatitis, current alcohol abuse, or cirrhosis.
26. Autoimmune disease requiring immunosuppressive therapy, except for up to 10 mg prednisone daily (or equivalent).
27. Seizure disorder requiring therapy within the past 12 months. Subjects with a history of seizure disorder beyond must have a complete CNS workup.
28. Major surgery within 4 weeks of the first dose of study drugs, except for lymphoma reasons.
29. Any other co-existing medical or psychological condition that will preclude participation in the study or compromise the ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Best overall response rate (BORR) | 12 months after the start of study therapy
  BORR defined as the proportion of patients with r/r DLBCL, HGBL and FL grade 3B who achieve a complete or partial remission as best response up to 12-months of study treatment according to the 2014 Lugano criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years after the start of study therapy
  2-year progression-free survival (PFS) with a 95% confidence interval. PFS is defined as time from the first dose of study drug until one of the following events occurs, whichever is first: Disease progression, Relapse or Death due to any cause. Patients who have not experienced an event at the time of analysis will be censored at the most recent date of disease assessment.
Overall survival (OS) | 2 years after the start of study therapy
  2-year overall survival (OS) defined as the time from the first dose of study drug to death of any cause. Patients who have not experienced an event at the time of analysis will be censored at the last date known to be alive.
Complete response (CR) rate | 12 months after the start of study therapy
  Complete response (CR) rate measured as the number of complete remissions as best response (achieved up to 12 months) divided by the number of patients treated with at least one dose of study drug.
Partial response (PR) rate | 12 months after the start of study therapy
  Partial response (PR) rate measured as the number of partial remissions as best response (achieved up to 12 months) divided by the number of patients treated with at least one dose of study drug.
Time to complete response | from the start of therapy to documentation of complete remission
  Time to complete response measured as the time from the start of therapy to documentation of complete remission.
Time to best response | 12 months after the start of study therapy
  Time to best response (achieved up to 12 months) measured as the time from the start of therapy to documentation of the best tumor response according to type of response.
Duration of response | from documentation of tumor response (complete or partial remission) to relapse or progressive disease
  Duration of response measured as the time from documentation of tumor response (complete or partial remission) to relapse or progressive disease.
BORR after 18-months of treatment | 18 months after the start of study therapy
  BORR defined as the best overall response of complete or partial remission after 18-months of treatment.
BORR after 24-months of treatment | 24 months after the start of study therapy
  BORR defined as the best overall response of complete or partial remission after 24-months of treatment.
Progression rate | 12 months after the start of study therapy
  Progression rate measured as the number of progressions (observed up to 12 months) divided by the number of patients treated with at least one dose of study drug.
Rate of relapse | From date of complete or partial remission until the date of relapse, assessed until the end of the study
  Relapse rate measured as the number of relapses divided by the number of patients included with complete or partial remission.
Biological characteristics of the lymphoma | Screening visit (day -28 to day -1); during therapy cycles of loncastuximab tesirine and epcoritamab; end of trial, or in case of relapse/progression, or subject discontinuation, whichever comes first.
  Outcomes of the study will be evaluated according to biological characteristics of the lymphoma.
Adverse Events (AEs) | AEs will be assessed at each study visit from start of the study until 150 days after the last administration of loncastuximab tesirine and/or epcoritamab (whichever is administered last).
  AEs that occurred in the study.
Serious Adverse Events (SAEs) | SAEs will be assessed at each study visit from start of the study until 150 days after the last administration of loncastuximab tesirine and/or epcoritamab (whichever is administered last).
  SAEs that occurred in the study.
Rate of treatment-related deaths | from start of the therapy to 2 months after the end of therapy
  Rate of treatment-related deaths defined as the number of treatment-related deaths during therapy or up to 2 months after the end of therapy divided by the number of patients treated with at least one dose of study drug.
Number and duration of treatment cycles and cumulative doses of loncastuximab tesirine and epcoritamab | At each therapy cycle from start of the study therapy until the last administration of loncastuximab tesirine and/or epcoritamab (whichever is administered last).
  Number of treatment cycles received, duration of treatment cycles and cumulative doses of loncastuximab tesirine and epcoritamab.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Münster, Medizinische Klinik A, Münster, Germany

IPD SHARING:
Plan to Share IPD: No